CLINICAL TRIAL: NCT00571116
Title: Evaluation of Disulfiram Plus Arsenic Trioxide In Patients With Metastatic Melanoma and at Least One Prior Systemic Therapy (Phase 1b)
Brief Title: Disulfiram Plus Arsenic Trioxide In Patients With Metastatic Melanoma and at Least One Prior Systemic Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Halted because of slow accrual and lack of study funding
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, John P. Fruehauf, Associate Clinical Professor of Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 06-08; 2006-5033 (Other: University of California, Irvine); NCI-2010-00338 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2007-12-06; First posted 2007-12-11 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic Melanoma; Disulfiram; Arsenic Trioxide; Metastatic Melanoma and at Least One Prior Systemic Therapy
MeSH Terms: conditions — Melanoma | interventions — Disulfiram; Arsenic Trioxide; arsenous acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Disulfiram and arsenic trioxide (Experimental): Patients receive disulfiram 250 mg PO twice daily and arsenic trioxide IV over 1-2 hours on Monday through Friday, alternating two weeks on treatment followed by two weeks off treatment. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.
  The Arsenic trioxide dose will be escalated or reduced until a tolerable dose is reached. Arsenic trioxide will be administered at a starting dose of 0.05 mg/kg. If the initial dose is tolerated, the patient will be dose escalated to 0.10 mg/kg/day. If the first dose escalation is tolerated, then a second dose escalation will be attempted to 0.15 mg/kg/day, the current dose recommended for leukemia. Dosing will be continued for two weeks on alternating with two weeks off as long as tolerated to a maximum of 60 doses.
  Interventions: Drug: Disulfiram; Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Disulfiram — Given PO
  Other Names: Antabuse; 25953; 97-77-8; bis(diethylthiocarbamoyl) disulfide; DS; tetraethylthioperoxydicarbonic diamide; tetraethylthiuram disulfide; Teturamin; TTD
Drug: Arsenic trioxide — Given IV
  Other Names: TRISENOX; 1327-53-3; 57974; 706363; Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid; Arsenous Acid Anhydride; Arsenous Oxide; AS2O3; White Arsenic

SUMMARY:
This phase I trial is studying the side effects and best dose of arsenic trioxide when given together with disulfiram in treating patients with metastatic and progressive melanoma. Drugs used in chemotherapy, such as disulfiram and arsenic trioxide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the tolerability of disulfiram and arsenic trioxide administration as a therapeutic combination. (Phase IB)

SECONDARY OBJECTIVES:

l. Determine the response rate (complete and partial responses) and time to progression of previously treated patients with metastatic malignant melanoma when treated with disulfiram plus Arsenic Trioxide. (Phase II)

OUTLINE: This is a dose-escalation study of arsenic trioxide.

Patients receive disulfiram orally (PO) twice daily and arsenic trioxide intravenously (IV) over 1-2 hours on Monday through Friday, alternating two weeks on treatment followed by two weeks off treatment. Courses repeat every 12 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have bidimensionally measurable disease. All measurable lesions must be assessed (by physical examination, CT scan, radionuclide scan or plain X-ray) within 28 days prior to registration. Non-measurable sites must be assessed within 42 days prior to registration. The subject's disease status must be completely assessed and reported.
* All subjects must undergo a CT of abdomen and chest within 28 days prior to registration.
* All subjects must undergo either a CT or MRI of the brain within 28 days of registration. Subjects with asymptomatic brain metastasis are eligible for this protocol but their metastasis must be clinically stable and asymptomatic. Subjects with Central Nervous System (CNS) metastasis must have been evaluated by neurosurgery prior to entry to confirm that they are a candidate for this trial. Treatment of symptomatic CNS metastasis that is required before protocol entry.
* Subjects must have progressed based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria after at least one prior systemic therapy (chemotherapy, biologic/immunotherapy, or a combination regimen) for metastatic disease. This includes development of any new lesion or a 20% increase in the sum of the subject's measurable disease compared to their previous nadir. New CNS metastasis could be the reason for disease progression, but they must be stable clinically and satisfy criteria delineated in section 5.4. Prior systemic therapy must have been completed at least 28 days before registration.
* Subjects may have received prior biologic or immunotherapy given in an adjuvant fashion. Prior adjuvant therapy must have been completed at least 28 days prior to registration
* Subjects may have received prior radiation therapy. If all known sites of disease have been previously radiated, there must be objective evidence of progression for the subject to be eligible. Radiation therapy must have been completed at least 28 days before registration.
* Subjects may have received prior surgery. Prior surgery must have been completed at least 28 days before registration.
* Performance status must be 0-2 according to Southwest Oncology Group Criteria

Performance Status:

GRADE SCALE

0 Fully active; able to carry on all pre-disease activities without restriction.

1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
2. Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours.
3. Capable of only limited self care; confined to bed or chair more than 50% of waking hours.
4. Completely disabled. Cannot carry on any self care. Totally confined to bed or chair.
5. Dead

   * Subjects must have a normal ECG, without evidence of congestive heart failure.

     1. Normal heart rate (less than 100 per minute)
     2. Normal sinus rhythm
     3. Normal interval from the beginning of the Q wave to the termination of the S wave, representing the time for ventricular depolarization (QRS) interval
     4. Subjects with QT prolongation > 500msec on their ECG will be considered ineligible.

        Exclusion Criteria:
   * Pregnant or nursing women are not eligible to participate in this trial because the safe use of this drug in pregnancy has not been established.
   * Subjects with severe myocardial disease or coronary occlusion, psychoses, and hypersensitivity to disulfiram or other thiuram derivatives used in pesticides and rubber vulcanization are excluded from the study.
   * Subjects who can not abstain from alcohol intake during the entire duration of this protocol are not qualified for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: Identification of Maximum Tolerated Dose | Up to 6 years
  The dose will be escalated or reduced until a tolerable dose is reached. Dose toleration is determined by the absence of any grade III/IV toxicities. Arsenic trioxide will be administered intravenously at a starting dose of 0.05 mg/kg daily, 5 days per week, for 2 weeks. The patients then have 2 weeks off, followed by two weeks of daily administration. If the initial dose is tolerated, the patient will be dose escalated for the second two weeks of drug administration to 0.10 mg/kg/day for two additional weeks, followed by two weeks off. If the first dose escalation is tolerated, then a second dose escalation will be attempted to 0.15 mg/kg/day, the current dose recommended for leukemia. The 0.15 mg/kg/day dose will be continued for two weeks on alternating with two weeks off as long as this is tolerated to a maximum of 60 doses. For patients developing grade III/IV toxicity at a given dose level, they will be dose reduced by one level and remain on that dose for the trial.

SECONDARY OUTCOMES:
Response rate (complete or partial response) | Up to 6 years
  Will be calculated as percentage of the study population. Data will be summarized in tabular form for publication.

CONTACTS AND LOCATIONS:
Overall Officials: John P Fruehauf, M.D. PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California, Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No